CLINICAL TRIAL: NCT06415812
Title: Evolutionary Systems Therapy for Early Onset of Personality Pathology: A Pilot Study on the Effectiveness and Feasibility With Adolescents and Young Adults
Brief Title: Evolutionary Systems Therapy for Personality Pathology
Acronym: ESTP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tages Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0124
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Personality Disorders
Keywords: compassion; metacognition; personality disorder; personality pathology; evolutionary psychopathology
MeSH Terms: conditions — Personality Disorders

STUDY DESIGN:
Intervention Model Description: Two individual parallel groups will be recruited: adolescent patients and young adult patients. Both groups will receive a 6-month Evolutionary Systems Therapy treatment. Both groups will access a longitudinal evaluation of the effectiveness of the treatment. All the participants will access a more extensive ecological momentary assessment to evaluate the progress of specific psychopathological mechanisms that are the targets of the treatment. Consistent with the conceptualization model of Evolutionary Systems Therapy and with the scientific literature on dimensional and hierarchical models of psychopathology, this conceptualization will be shared with the patient based on three macro-functionings: externalizing patterns, internalizing patterns, schizotypal patterns.
Masking Description: All data will be collected in a blinded manner by an assessor other than the therapists. Subsequently, the data will be anonymized and analyzed by a researcher from an institution different from the one in which the study takes place.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychotherapy (Experimental): All the participants receive as active treatment a form of psychotherapy for personality disorders (Evolutionary Systems Therapy). The treatment last 6 months (24 weekly sessions, each lasting 50-60 minutes).
  Interventions: Behavioral: Evolutionary Systems Therapy

INTERVENTIONS:
Behavioral: Evolutionary Systems Therapy — Evolutionary Systems Therapy is an individual form of psychotherapy (talk therapy) that has been previously tested trough a randomized controlled trial and a few cases series, confirming its feasibility and safety.

SUMMARY:
Evolutionary Systems Therapy is a new form of therapy that has been previously tested in a randomized controlled trial and in a few cases of patients diagnosed with Cluster A personality disorders. The objective of the present study is to investigate the feasibility and preliminary efficacy of Evolutionary Systems Therapy in all forms of personality disorders. The study includes three project actions: (i) a case series on adolescents with personality disorders; (ii) a case series on young adults with personality disorders; (iii) an ecological momentary assessment study to confirm the conceptualization model on all the patients.

DETAILED DESCRIPTION:
To explore the feasibility and preliminary efficacy of Evolutionary Systems Therapy, the present study includes three actions. In the first action investigators enroll 6 adolescents (16-19 years) with personality disorders, in the second 15 young adults (20-25 years) with personality disorders. All participants receive 6 months of psychotherapy. The two subsamples of patients (adolescents and young adults) are assessed based on the conceptualization model of Evolutionary Systems Therapy which envisages three macro-organizations of personality (consistently with dimensional and hierarchical models such as Hierarchical Taxonomy of Psychopathology): internalizing, externalizing, schizotypal. Investigators plan to recruit patients until the size of the sub-samples is reached (15 young adults divided into 3 groups of 5 patients, each for each of the three interpersonal patterns; 6 adolescents divided into 3 groups of 2 patients, each for each of the three patterns interpersonal). In the third action, an ecological momentary assessment study will investigate the consistency over time between the conceptualization model and the experiences of the young adult patients enrolled: investigators will explore whether the hypothesized conceptualization will be confirmed by collected data on the patients' interpersonal styles.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with personality pathology in accordance with Structured Clinical Interview for DSM-5 - Alternative Model of Personality Disorders Module I
* Being capable of read and sign the inform consent form

Exclusion Criteria:

* Being diagnosed with schizophrenia spectrum disorders and other psychosis
* Being diagnosed with bipolar disorders
* Being diagnosed with autism spectrum disorder
* Being diagnosed with intellectual disability
* Being under any psychopharmacological or psychosocial treatment

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Rate of individual change in personality pathology over time | 9 measurements: one month before the start of therapy, at the start of therapy, at the end of each of the 6 months of therapy, one month after the end of therapy.
  At least 75% rate of change in personality pathology over time as defined by a downward trend in mean of total score of Personality Inventory for DSM-5 Brief Form)
Group change in personality pathology over time | 9 measurements: one month before the start of therapy, at the start of therapy, at the end of each of the 6 months of therapy, one month after the end of therapy.
  Group change in personality pathology over time as defined by statistically significant change of sample mean of total score of Personality Inventory for DSM-5 Brief Form)
Feasibility of the intervention | 6 measurements: at the end of each of the six months of therapy
  At least 70% rate of completion, adherence, therapeutic alliance and adverse events

SECONDARY OUTCOMES:
Differential effect of the intervention between interpersonal patterns | 9 measurements: one month before the start of therapy, at the start of therapy, at the end of each of the 6 months of therapy, one month after the end of therapy.
  Comparison between efficacy of intervention between three interpersonal patterns (internalizing, antagonistic, schizotypal) as being the target of the intervention. The comparison is aimed to show no statistically significant difference between the three patterns in terms of pre-post change in personality pathology as measured by Personality Inventory for DSM-5 Brief Form
Specific effect of the intervention between interpersonal patterns | 40 measurements: 20 measurements in the month before surgery (2 measurements per day for the 10 days before the start of therapy) and 20 measurements in the month after surgery (2 measurements per day for the 10 days after the end of therapy)
  Comparison between efficacy of intervention between three interpersonal patterns (internalizing, antagonistic, schizotypal) as being the target of the intervention. The comparison is aimed to show no statistically significant difference between the three patterns in terms of pre-post change in personality pathology as measured by Personality Inventory for DSM-5 Brief Form.
Remission from diagnosis | 2 measurements: one at baseline assessment (once the intervention starts); one at final assessment (6 months after, that is after weekly scheduled 24 sessions)
  At least 70% rate of remission from diagnosis of personality pathology

CONTACTS AND LOCATIONS:
Overall Officials: Simone Cheli, PhD, Principal Investigator — Tages Onlus
Locations (1):
- Centro di Psicologia e Psicoterapia Tages Onlus - Firenze, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: Yes
All the data collected as well as the study documents will be available on the Open Science Foundation no later than September 2024
Supporting Information: Study Protocol, SAP, ICF
Time Frame: May 2024
Access Criteria: Open Access
URL: https://osf.io/urjdz/

REFERENCES:
- [Background] Cheli, S., Chiarello, F., & Cavalletti, V. (2023). A psychotherapy oriented by compassion and metacognition for schizoid personality disorder: A two cases series. Journal of Contemporary Psychotherapy: On the Cutting Edge of Modern Developments in Psychotherapy, 53(1), 61-70. https://doi.org/10.1007/s10879-022-09566-3
- [Background] Cheli, S., Cavalletti, V. An Evolutionarily Oriented Therapy for Autistic Adolescents with Extraordinary Skills: A Two-Case Series. J Contemp Psychother 53, 297-304 (2023). https://doi.org/10.1007/s10879-023-09586-7
- [Background] Cheli, S., & Brüne, M. (In press). When do personality traits become pathological? An epistemological and evolutionary view. To appear in Konrad Banicki and Peter Zachar (Eds.), Novel Conceptual Approaches to Personality Disorders for Psychologists and Philosophers. Cambridge University Press.
- [Result] Cheli S, Cavalletti V, Lysaker PH, Dimaggio G, Petrocchi N, Chiarello F, Enzo C, Velicogna F, Mancini F, Goldzweig G. A pilot randomized controlled trial comparing a novel compassion and metacognition approach for schizotypal personality disorder with a combination of cognitive therapy and psychopharmacological treatment. BMC Psychiatry. 2023 Feb 20;23(1):113. doi: 10.1186/s12888-023-04610-5. PMID 36803673
- [Result] Cheli S, Goldzweig G, Chiarello F, Cavalletti V. Evolutionary systems therapy for paranoid personality disorder: A seven cases series. Bull Menninger Clin. 2024 Winter;88(1):61-80. doi: 10.1521/bumc.2024.88.1.61. PMID 38527104